CLINICAL TRIAL: NCT01077479
Title: Metformin in Preventing Androgen Deprivation Therapy Induced Insulin Resistance and Metabolic Syndrome
Acronym: MVENT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Western Sydney Local Health District (Other)
Responsible Party: Principal Investigator, Howard Gurney, A/Prof Howard Gurney, Western Sydney Local Health District
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: HGWH009
Record Dates: First submitted 2010-02-26; First posted 2010-03-01 (Estimated); Last update posted 2014-05-15 (Estimated); Status verified 2014-05

CONDITIONS: Metabolic Syndrome; Hypercholesterolemia
Keywords: body fat mass gain; Insulin resistance
MeSH Terms: conditions — Metabolic Syndrome; Hypercholesterolemia; Insulin Resistance | interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Metformin (Experimental)
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Metformin — Metformin 1500mg nocte for 6 months

SUMMARY:
The main purpose of this study is to assess the efficacy of metformin in abrogating androgen deprivation therapy (ADT) induced insulin resistance as measured by homeostasis model assessment (HOMAIR) in men with non-metastatic prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age
* ECOG ≤ 1
* Histologically confirmed prostate cancer of early or locally advanced stage, or metastatic prostate cancer with bone involvement only (≤ 5 sites of bone metastases only)
* Plan to receive ≥ 6 months continuous androgen deprivation therapy by a GnRH agonist
* Patients who are to receive antiandrogens with GnRH agonists are not excluded from the study. But the form, dose and duration of antiandrogen treatment should be recorded.
* Adequate renal function (Creatinine ≤ 177mMol/L and GFR >30 mls/min )
* Adequate hepatic function (Bilirubin must be ≤ 1.5 x upper limit of normal range, ALT and ALP must be ≤ 2.5 x upper limit of normal)

Exclusion Criteria:

* Visceral involvement
* > 5 sites of bone metastases
* History of confirmed diabetes mellitus (patients with impaired fasting glucose or impaired glucose intolerance will not be excluded) 12
* Treatment with medications that may alter glucose or insulin level within 3 months (including insulin, oral hypoglycemic agents, systemic corticosteroid of any dosage, atypical antipsychotic drugs of any dose)
* Malignant disease other than prostate cancer at the time of enrolment
* Bilateral orchiectomy
* Previous androgen deprivation therapy by a GnRH agonist or anti-androgen within last 12 months(patient who had a GnRH agonist more than 12 months ago are allowed if their testosterone levels are in the normal range at the time of recruitment)
* Chemotherapy within 6 months
* History of lactic acidosis
* Cardiac or respiratory insufficiency, severe infection that is likely to increase the risk of lactic acidosis
* Medical or psychiatric conditions that compromise the patient's ability to give informed consent

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2010-02; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
The percentage change in insulin resistance measured by homeostasis model assessment (HOMAIR) from baseline to 12 and 24 weeks | 12 and 24 weeks

SECONDARY OUTCOMES:
To assess the efficacy of metformin in abrogating ADT-induced insulin resistance as measured by whole-body insulin sensitivity index(ISI) at 3 and 6 months | 12 and 24 weeks
To assess the efficacy of metformin in reducing the incidence of ADT-induced metabolic syndrome at 3 and 6 months | 12 and 24 weeks
To assess the efficacy of metformin in reducing ADT-induced percentage body fat mass gain 6 months | 24 weeks
To assess the efficacy of metformin in reducing ADT-induced hypercholesterolemia at 3 and 6 months | 12 and 24 weeks
To validate measurement of insulin resistance by HOMAIR with euglycemic hyperinsulinemic clamp in a subgroup group of participants | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Howard Gurney, MBBS, FRACP, Principal Investigator — Westmead Cancer Care Centre
Locations (1):
- Westmead Hospital, Sydney, New South Wales, Australia